CLINICAL TRIAL: NCT03712696
Title: A Study on the Efficacy and Safety of DIGNICAP™ System for Preventing Chemotherapy Induced Alopecia
Brief Title: Efficacy and Safety of DIGNICAP™ System
Acronym: DIGNICAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IEO 0075/
Record Dates: First submitted 2018-09-25; First posted 2018-10-19 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Breast Cancer; Chemotherapy-induced Alopecia
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DIGNICAP™ (Experimental): DigniCap® System
  Interventions: Device: DIGNICAP™

INTERVENTIONS:
Device: DIGNICAP™ — Scalp cooling to prevent chemotherapy-induced alopecia

SUMMARY:
Chemotherapy-induced alopecia (CIA) is one of the most common and emotionally distressing side effects of cancer therapy.

In this study we sought to assess the feasibility and the effectiveness of scalp cooling system DigniCap® to prevent alopecia in primary breast cancer patients receiving an anthracycline containing adjuvant chemotherapy (CT).

A prospective two-stage design clinical trial conducted at a single Institution of women with primary breast cancer scheduled to receive anthracycline with or without taxane-based adjuvant CT. Patients were enrolled from July 2014 to November 2016, with ongoing annual follow up for 5 years.

The scalp cooling period initiated approximately 30 minutes before CT. Scalp temperature was to be maintained at 3-5°C throughout CT and for 90 to 120 minutes afterward, depending on the CT drug and dose.

DETAILED DESCRIPTION:
Scalp cooling to prevent chemotherapy-induced alopecia has been in use since the 1970's and offers excellent or good prevention of alopecia caused by many chemotherapeutic regimens, including those commonly used for breast cancer. The protection from alopecia offered by scalp cooling is a consequence of vasoconstriction resulting in reduced blood flow in the scalp, and reduced metabolic rate in the hair follicles with consequent decreased exposure to the chemotherapeutic agents. This limits the damage to dividing cells in the hair follicles.

In general, scalp cooling is well tolerated. Tolerance can be graded by a Visual Analogue Scale of 0-10, in which 0 represents 'not tolerable' and 10 means 'really well tolerable'. Mean scores vary between 6.9 and 8.0. No serious side effects have been reported. The most common reported side effects are headaches, unpleasant feelings due to the heaviness of the cap and coldness, dizziness and transient lightheadedness. Headaches are mostly not severe and can usually be prevented by paracetamol. Freezing has never been reported. Side effects in more than 10% of the patients were the reason to stop scalp cooling in only four of all studies.

DigniCap® System has been developed to provide continuous scalp cooling with high efficacy, safety and acceptable patient comfort. The system consists of a refrigerator unit integrated into a control unit based on a computerized interface. The system forms a compact mobile cabinet to which a soft and tight-fitting silicon cap is connected via a tube. A liquid coolant is pumped from the cooled reservoir in the cabinet to circulate through small canals within the cap. Two separate cooling circuits allow coolant to flow through the front and the back of the cap autonomously. Scalp temperature is monitored by three separate sensors in the cap: two temperature sensors and a security sensor. Deviations from the preset temperatures are immediately detected and automatically adjusted by the system. An outer cap made of neoprene is used to secure and insulate the inner silicon cap.

Since hair loss becomes noticeably visible after the loss of 50% or more of the scalp hair, the efficacy and safety of the Dignicap System to prevent chemotherapy induced alopecia will be evaluated in women with early breast cancer undergoing adjuvant chemotherapy regimens. The scalp cold cap will be applied at each chemotherapy cycle. Hair loss will be evaluated by patient self assessment (VAS scale), and by means of 5 standardized photographs taken prior to each chemotherapy cycle and by physician by the 5 point Dean's scale.

ELIGIBILITY:
Inclusion Criteria:

* Women > 18 years of age Performance status (ECOG) 0- 1
* Documented diagnosis of stage I or II breast cancer
* A planned course of chemotherapy in the adjuvant setting with curative intent including one of the following regimens:

  * Doxorubicin 60 mg/m2 or Epirubicin 90 mg/m2 and cyclophosphamide 600 mg/m2 x 4 cycles IV every 3 weeks
  * Docetaxel 75 mg/m2 and cyclophosphamide 600 mg/m2 x 4 cycles IV every 3 weeks
  * Paclitaxel 80 mg/m2 weekly IV x at least 12 weeks with or without IV trastuzumab
  * Docetaxel 75-100 mg/m2 IV every 3 weeks x 4 cycles with or without trastuzumab IV weekly or every 3 weeks
  * Targeted agents such as trastuzumab are allowed
  * Patients receiving a regimen including both an anthracycline and a taxane (at doses reported above) are also eligible for this trial (AC/T, EC/T, TAC, etc.)
* Plan to complete chemotherapy within 6 months
* Willing and able to sign informed consent for protocol treatment
* Willing to participate in study procedures including having photographs of the head before the first cycle of chemotherapy and 1 month after the last chemotherapy
* Willing to enroll in an extension protocol for follow up for 5 years following the end of chemotherapy treatment
* Negative pregnancy test (in fertile women).

Exclusion Criteria:

* Patients with female pattern baldness resembling picture I-3 or higher on the Savin scale
* Previous chemotherapy
* Autoimmune disease affecting hair; e.g. alopecia areata, systemic lupus with associated hair loss
* A history of whole brain radiation
* Plans to use a chemotherapy regimen other than those specified in the inclusion criteria.
* Concurrent hormone therapy with chemotherapy except LHRH analogue. Hormone therapy should be used as indicated following completion of chemotherapy
* Underlying clinically significant liver disease including active viral hepatitis with abnormal liver function tests >1.5 times the upper limit of normal, including alkaline phosphatase, AST, and total bilirubin. Patients with Gilbert´s disease (elevated indirect bilirubin only) will be eligible for participation.
* Clinically significant renal dysfunction defined as serum creatinine > upper limit of normal.
* A serious concurrent infection or medical illness which would jeopardize the ability of the patient to complete the planned therapy and follow-up
* A history of persistent grade 2 (or higher) alopecia induced by prior chemotherapeutic regimens
* Participation in any other clinical investigation or exposure to other investigational agents, drugs, device or procedure that may cause hair loss Intercurrent life-threatening malignancy
* A history of cold agglutinin disease or cryoglobulinemia.
* Evidence of untreated or poorly controlled hyper or hypothyroidism
* A history of silicon allergy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2014-07-18 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-09-20 (Actual)

PRIMARY OUTCOMES:
Reduction of hair loss | 21 days
  Hair loss (HR) assessed by the patient herself after completing the last cycle of chemotherapy (21 days after last CT infusion) using photographs taken 5 angles using a VAS (Visual Analogue Scale) (Grade 0: no hair loss; Grade 1: < 25% hair loss; Grade 2: 25-50% of hair loss; Grade 3: 50-75% of hair loss; Grade 4: >75% of hair loss)

SECONDARY OUTCOMES:
Hair loss assessed by physician | 21 days
  Reduction of hair loss assessed by physician by the 5 point Dean's scale (Judith C Dean's Scale for hair loss) (Grade 0: no hair loss; Grade 1: < 25% hair loss; Grade 2: 25-50% of hair loss; Grade 3: 50-75% of hair loss; Grade 4: >75% of hair loss)
Assessment of head/scalp pain | 21 days
  Assessment of head/scalp pain using a Visual Analogue Scale (VAS) from 0 (not tolerable) to 100 (really well tolerable)
Assessment of feeling chilled | 21 days
  Assessment of feeling chilled using a Visual Analogue Scale (VAS) from 0 (not at all chilled) to 10 (as bad as it could be)
Assessment of patient satisfaction | 21 days
  Assessment of patient satisfaction using Technology Acceptance Model Questionnaire
Assessment of patient symptoms | 21 days
  Assessment of patient symptoms using EORTC QLQ BR-23 Questionnaire
Assessment of patient health status | 21 Days
  Assessment of patient health status using EORTC QLQ C-30 Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Elisabetta Munzone, MD, Principal Investigator — IEO
Locations (1):
- European Institute of Oncology, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Munzone E, Bagnardi V, Campenni G, Mazzocco K, Pagan E, Tramacere A, Masiero M, Iorfida M, Mazza M, Montagna E, Cancello G, Bianco N, Palazzo A, Cardillo A, Dellapasqua S, Sangalli C, Pettini G, Pravettoni G, Colleoni M, Veronesi P. Preventing chemotherapy-induced alopecia: a prospective clinical trial on the efficacy and safety of a scalp-cooling system in early breast cancer patients treated with anthracyclines. Br J Cancer. 2019 Aug;121(4):325-331. doi: 10.1038/s41416-019-0520-8. Epub 2019 Jul 15. PMID 31303642